CLINICAL TRIAL: NCT02027116
Title: Multi-center, Open-label, Dose Escalation, Phase I Trial to Evaluate the Safety, Tolerability and Immunogenicity of VGX-6150 for Second-line Therapy of Chronic Hepatitis C Infection
Brief Title: Phase I Trial to Evaluate the Safety, Tolerability and Immunogenicity of VGX-6150 for Second-line Therapy of Chronic Hepatitis C Infection
Acronym: VGX-6150-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGX-6150-01
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C; DNA Vaccine; Electroporation; Intramuscular (IM) Injection
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: 1mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-6150 containing 1mg DNA/dose administered via IM injection + electroporation at Day 0, Week 4, Week 8, Week 12
  Interventions: Biological: VGX-6150
- Experimental: 3mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-6150 containing 3mg DNA/dose administered via IM injection + electroporation at Day 0, Week 4, Week 8, Week 12
  Interventions: Biological: VGX-6150
- Experimental: 6mg of DNA/dose (Experimental): Subjects will receive a 3 dose series of VGX-6150 containing 6mg DNA/dose administered via IM injection + electroporation at Day 0, Week 4, Week 8, Week 12
  Interventions: Biological: VGX-6150

INTERVENTIONS:
Biological: VGX-6150 — Plasmid DNA delivered via IM injection with electroporation

SUMMARY:
To evaluate the safety, tolerability and immunogenicity of VGX-6150 as second-line therapy in chronic hepatitis C patients

ELIGIBILITY:
Inclusion Criteria:

* Subjects who want to participate in this trial should meet all of the following criteria.

  1. Male or females aged 19 to 65 years
  2. Chronic hepatitis C patients infected with HCV genotype 1a or 1b
  3. Patients who failed* SOC therapy with PEG-IFN and ribavirin or triple therapy with SOC and DAA agents

     *Treatment failure is defined by any of the following; A. Partial response (PR) Serum HCV RNA level declined by at least 2 log10 but still detected at treatment week 24 B. Non-response (NR) Serum HCV RNA level not declined by at least 2 log10 at treatment week 12 C. Relapse Serum HCV RNA undetected during treatment but detectable after end of treatment D. Treatment discontinuation due to ADR or other reason
  4. Patients whose deltoid muscles (left or right) are accessible by 12 to 19 mm cannula/ electrode for intramuscular (IM) injection and electroporation (EP)
  5. Patients who can comply with planned schedule of this protocol
  6. Patients who give written informed consent voluntarily

Exclusion Criteria:

* Subjects who meet any of the followings cannot participate in this study.

  1. Liver transplant recipients
  2. Patients having decompensated liver cirrhosis with any history or evidence of ascites, esophageal variceal hemorrhage and/or hepatic encephalopathy
  3. Malignant tumor patients who received radiotherapy or chemotherapy before study participation
  4. Current active infection except hepatitis C that requires medical treatment
  5. Autoimmune disease patients or immunodeficient (immuno-compromised) patients
  6. Patients who received immunomodulators, cytotoxic agents or systemic corticosteroids for chronic disease other than hepatitis C within 2 months before study participation
  7. Patients who received non-steroidal anti-inflammatory drugs (NSAIDs) within 10 days before IP administration
  8. Concomitant diseases which is judged to be unacceptable for study participation by investigator (e.g., severe cardiovascular, renal , or psychiatric disease)
  9. Clinically significant abnormal findings in physical examination,laboratory tests, vital signs or ECG at investigator's discretion
  10. Patients with implantable pacemaker
  11. Patients with metal implant in IP administration area or nearby
  12. Positive for HBsAg, or HIV Ab
  13. Previous history of gene therapy
  14. History of allergy or anaphylaxis to any component of IP or other vaccine
  15. Patients who received major surgery within 4 weeks before IP administration
  16. Blood transfusion within 4 weeks before IP administration
  17. Current alcohol or drug abuse
  18. Patients who received other vaccine within 30 days before IP administration
  19. Pregnancy or breast-feeding woman
  20. Women of childbearing potential (WOCBP) or men with partner of WOCBP who are unwilling to use adequate contraception or be abstinent during the trial
  21. Patients who received other investigational products within 30 days before study participation
  22. Patients incapable of participating in this trial by investigator's judgment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Screening ~ week 36
  To evaluate the safety and tolerability of VGX-6150 as second-line therapy in chronic hepatitis C patients.

SECONDARY OUTCOMES:
Immunogenicity and virologic response | Screening ~ Week 36
  To evaluate the immunogenicity and virologic response to VGX-6150 in treatment failure patients with chronic hepatitis C

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, M.D, Ph.D., Principal Investigator — Severance Hospital; Jeong Heo, M.D, Ph.D., Principal Investigator — Pusan National University Hospital
Locations (2):
- South Korea (2):
  - Pusan National University Hospital, Pusan
  - Yonsei University Severance Hospital, Seoul

REFERENCES:
- [Derived] Han JW, Sung PS, Hong SH, Lee H, Koh JY, Lee H, White S, Maslow JN, Weiner DB, Park SH, Jeong M, Heo J, Ahn SH, Shin EC. IFNL3-adjuvanted HCV DNA vaccine reduces regulatory T cell frequency and increases virus-specific T cell responses. J Hepatol. 2020 Jul;73(1):72-83. doi: 10.1016/j.jhep.2020.02.009. Epub 2020 Feb 21. PMID 32088322